CLINICAL TRIAL: NCT04659252
Title: Circulating Tumour Protein Quantification From Capillary Blood for Patient Selfsampling and Safe Remote Monitoring of Multiple Myeloma During COVID-19
Brief Title: CORONADO (Circulating tumOur pROtein quaNtification cApillary blooD cOvid-19)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR5361
Record Dates: First submitted 2020-12-08; First posted 2020-12-09 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: n/a - samples collected along routine care samples only — This is a non-interventional study.

SUMMARY:
The coronavirus (COVID-19) pandemic has brought severe challenges for myeloma patients. Myeloma patients are considered ultra-high risk for COVID-19 and fall into the strictest group for shielding. When on treatment, but also during times of active surveillance, patients have to regularly and frequently leave shielding and visit the hospital for blood tests to monitor their disese. This is specifically for quantification of circulating tumour protein biomarker tests for paraprotein (PP) and/or serum free light chains (sFLCs) by specialised biochemistry units.

This research aims to evaluate the potential use of an at-home patient administered technique to sample blood. The purpose of the blood sampling technique is to monitor your disease status. We want to test if it is possible to monitor a patient's disease status using this alternative blood collection method when compared to monitoring disease status using the traditional blood collection methods (venous blood sampling).

The new VAMS method is not intended to be used interchangeably or will not replace the current method. This study is to evaluate an alternative sample type that may be used to improve the patient pathway, especially during these uncertain times.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of a B-cell dyscrasia
2. Measurable disease by serum free light chain assay
3. Signed informed consent

Exclusion Criteria:

1. Patients <21 years of age
2. Cognitive impairment
3. Non-B Cell Dyscrasia patients

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multiple myeloma patients attending routine phlebotomy clinic.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2021-03-04 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Validated FLC | 6 months
  Validated FLC method for use with VAMS that conforms to ISO15189:2012 accreditation

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Boyd, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- The Royal Marsden NHS Foundation Trust, Sutton, United Kingdom

IPD SHARING:
Plan to Share IPD: No